CLINICAL TRIAL: NCT07259408
Title: Co-creation of Tools for People in Detention With Suicidal Thoughts and/or Behavior
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2025-0349
Record Dates: First submitted 2025-09-12; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Suicide Prevention; Suicide; Suicidal Ideation
Keywords: Safety Plan; Safety Planning; Suicide prevention; Risicoformulering; risk formulation; detention; prison; incarceration
MeSH Terms: conditions — Suicide Prevention; Suicide; Suicidal Ideation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals in detention: Participants are individuals in detention which is invited to participate in semi-structured interviews. If they agree, their referrer will schedule a date for the interview at the prison with the researcher.
  Interventions: Other: Co-creation process for suicide prevention tools in detention
- Professionals working in detention: Participants are professionals working in detention settings, such as psychologists, psychiatrists, social workers, and nurses. They are invited to participate in semi-structured interviews. If they agree, the researcher will contact them to schedule a date for the interview at the prison.
  Interventions: Other: Co-creation process for suicide prevention tools in detention

INTERVENTIONS:
Other: Co-creation process for suicide prevention tools in detention — The intervention consists of a co-creation process involving detained individuals and detention professionals through semi-structured interviews.
  For professionals, the interviews will focus on the usability, applicability, and implementation of three suicide prevention tools.
  Interviews with individuals in detention will focus only on the Safety Plan. They will be asked about what helps them in moments of crisis and their views on the Safety Plan in detention.
  The goal is to collect feedback on usability, perceived barriers, and suggestions for real-world implementation in the detention context. Interviews are repeated up to three times per professional participants depending on availability and co-creation progress. For individuals in detention there is only one interview. Feedback from all participants will be used to adapt and refine the tools for future use in detention facilities.

SUMMARY:
People in detention are at significantly higher risk of suicide compared to the general population. In Belgian prisons, the suicide rate is five times higher than average. Despite the availability of suicide prevention tools, many are not scientifically validated or adapted to the detention context, leading to inconsistent use and missed warning signs.

This study aims to evaluate and adapt three evidence-based suicide prevention tools-the Safety Plan, the guideline for the care and evaluation of suicidality , and the Risk Formulation template-for use in detention settings. Through interviews with both professionals working in prisons and individuals in detention, the study explores how these tools can be made more relevant, practical, and effective in this unique environment.

The research involves 40 participants: 20 professionals and 20 individuals in detention. Interviews will gather feedback on the tools' usability, clarity, and fit with the realities of prison life. The ultimate goal is to improve suicide prevention practices in detention by offering tailored, scientifically grounded tools that support both staff and detainees.

ELIGIBILITY:
For professionals working in detention:

Inclusion criteria:

* Aged 18 years or older
* Currently working in a professional care role within a prison setting (e.g., psychologist, psychiatirst, social worker, nurse, etc.)
* Experience in supporting or treating incarcerated individuals with suicidal thoughts or behaviours

Exclusion Criteria:

* Under the age of 18
* Not employed in a professional caregiving role within detention (e.g., correctional officers or security staff)

For people in detention:

Inclusion criteria:

* Aged 18 years or older
* Experienced suicidal thoughts within the past three years

Exclusion criteria:

* Under the age of 18
* Significant cognitive limitations that would make the participation in an interview infeasible
* Insufficient command of the Dutch language to understand and respond to interview questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from Belgian detention facilities and the prison-based care network. Specifically:
  * Professionals working in detention: Psychologists, psychiatrists, social workers, nurses, and other healthcare staff working within Belgian detention centers who have had experience in suicide prevention.
  * People in detention: Adults held in selected Belgian prisons who are clinically stable and able to participate in a one-hour interview. Referrals will be made by prison psychologists, social workers, or healthcare staff.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Suicide Prevention Tools in the Detention Context | Each participant is assessed during one (for incarcerated individuals) or up to three (for professionals) interviews
  This outcome measure assesses the usability, applicability, and improvement potential of three suicide prevention tools based on qualitative feedback from professionals working in detention and individuals in detention. Through semi-structured interviews, the study explores how these tools are experienced in practice, identifies perceived strengths and limitations, and gathers concrete suggestions for adaptation to better fit the detention environment.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — Flemish Centre of Expertise in Suicide Prevention (Ghent University)
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided